CLINICAL TRIAL: NCT00184301
Title: Treatment of Patients With Concurrent Eating Disorder and Personality Disorder: A Controlled Randomized Comparison Study, of Treatments Given to In-patients and Out-patients.
Brief Title: A Comparison Study of Treatments Given to Patients With Concurrent Eating Disorder and Personality Disorder.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other); Norwegian Foundation for Health and Rehabilitation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 064.03
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2017-03-29 (Actual); Status verified 2017-03

CONDITIONS: Eating Disorder; Anorexia Nervosa; Bulimia Nervosa; Personality Disorder
Keywords: Eating disorders; Anorexia nervosa; Bulimia nervosa; Personality disorders; In-patient treatment; out-patient treatment; group therapy
MeSH Terms: conditions — Feeding and Eating Disorders; Anorexia Nervosa; Bulimia Nervosa; Personality Disorders | interventions — Hospitalization; Ambulatory Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- inpatient treatment (Experimental): inpatient treatment during 1 year
  Interventions: Behavioral: inpatient treatment
- outpatient treatment (Active Comparator): intensive outpatient treatment consisting of two-weekly group sessions during 1 year
  Interventions: Behavioral: outpatient treatment

INTERVENTIONS:
Behavioral: inpatient treatment — inpatient treatment during 1 year
  Arms: inpatient treatment
Behavioral: outpatient treatment — intensive outpatient treatment consisting of two-weekly group sessions during 1 year
  Arms: outpatient treatment

SUMMARY:
The aim of this study is to determine whether in-patient treatment is better then intensive out-patient group treatment for patients with concurrent eating disorder and personality disorder.

DETAILED DESCRIPTION:
The main aim of the study is to compare the effects of in-patient treatment with a group based intensive out-patient treatment. It is a randomized controlled comparison study including patients with concurrent eating disorder and personality disorder. 18 patients will receive an in-patient treatment lasting one year. 18 patients will receive intensive out-patient treatment consisting of two-weekly group sessions, lasting one year. Personality disorder, eating behavior, symptoms, and function will be followed for two years.

ELIGIBILITY:
Inclusion Criteria:

* Anorexia nervosa, bulimia nervosa, personality disorder.

Exclusion Criteria:

* male, schizophrenia.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2005-09 (Actual); Primary Completion 2011-12 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Score on personality, interpersonal, eating disorder and symptom scales | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Are Holen, PhD MD, Principal Investigator — Norwegian University of Science and Technology
Locations (1):
- Østmarka Psychiatric Department, St Olavs Hospital, University Hospital of Trondheim., Trondheim, Norway

IPD SHARING:
Plan to Share IPD: No